CLINICAL TRIAL: NCT02486497
Title: Adjuvant Gemcitabine Versus 5-FU/Leucovorin Based on hENT1 Immunostaining After Curative Surgery of Pancreatic Cancer
Brief Title: Adjuvant Gemcitabine Versus 5-FU/Leucovorin Based on hENT1 Immunostaining
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: IlDong Pharmaceutical Co Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SNUBH-IMGPB-2015-01
Record Dates: First submitted 2015-06-23; First posted 2015-07-01 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2016-08

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic cancer; Adjuvant chemotherapy; hENT1; Gemcitabine
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 5-FU group (Active Comparator): Grades of hENT1 immunostaining are 0 or 1.
  Interventions: Biological: hENT1
- Gemcitabine group (Active Comparator): Grade of hENT1 immunostaining is 2.
  Interventions: Biological: hENT1

INTERVENTIONS:
Biological: hENT1 — hENT1 is a membrane transporter for gemcitabine. According to the hENT1 staining, patients will be treated with gemcitabine or 5-FU.

SUMMARY:
Human equilibrative nucleoside transporter 1 (hENT1) is a membrane transporter which is a predicting marker for gemcitabine chemotherapy. However, there is a limited evidence of it as an indicator for adjuvant gemcitabine chemotherapy. In this study, investigators try to investigate the role of hENT1 as a indicator of selection of adjuvant chemotherapy regimen between gemcitabine and 5-fluorouracil (5-FU).

DETAILED DESCRIPTION:
After surgical resection of pancreatic cancer, the tissue is immunostained by hENT1 antibody. The grades of immunostaining are categorized as 0 (0%), 1 (<50%), and 2 (>=50%). According to the grade, patients with grade 0 or 1 will be treated with 5-FU and those with grade 2 will be treated with gemcitabine. After the study, investigators will calculate the overall survival and recurrence free survival of the patients and investigate the role of hENT1 as a predictive biomarker for adjuvant gemcitabine chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with curatively resected pancreatic cancer
* Age between 18 and 75
* Eastern Cooperative Oncology Group performance score 0 or 1
* Patients with compliance
* Patients with informed consent

Exclusion Criteria:

* Patients refuse to enroll this study
* Patients with concomitant chemoradiation therapy
* Previous chemotherapy
* Pregnant or preparing a pregnancy
* Uncontrolled infection, diabetes, hypertension, ischemic heart disease, myocardial infarction within 6 months
* Enrolled another clinical trial within 30 days
* Patients will be expected to be risk because of enrollment
* Patients without informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-06; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Recurrence free survival | Upto 24 weeks

SECONDARY OUTCOMES:
Overall survival | Upto 24 weeks
Toxicity | Upto 24 weeks
  Hematologic and hepatic toxicity according to blood test results & non-hematologic toxicity (fatigue, vomiting, diarrhea, sensory neuropathy) according to CTCAE 4.0 scale

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Shin DW, Lee JC, Kim J, Yoon YS, Han HS, Kim H, Hwang JH. Tailored adjuvant gemcitabine versus 5-fluorouracil/folinic acid based on hENT1 immunohistochemical staining in resected pancreatic ductal adenocarcinoma: A biomarker stratified prospective trial. Pancreatology. 2021 Jun;21(4):796-804. doi: 10.1016/j.pan.2021.02.022. Epub 2021 Mar 4. PMID 33795193